CLINICAL TRIAL: NCT06958107
Title: Prospective Clinical Evaluation of Circulating Tumor DNA Liquid Biopsy in Sarcoma Patients
Brief Title: LCI-SAR-BSTS-CTDNA-001: Circulating Tumor DNA Liquid Biopsy in Sarcoma Patients
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Paula Takacs Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00127078; LCI-SAR-BSTS-CTDNA-001 (Other: Atrium Health)
Record Dates: First submitted 2025-04-27; First posted 2025-05-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Sarcoma
Keywords: circulating tumor DNA; liquid biopsy; bone or soft tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Alanine Transaminase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-Metastatic and Resectable: Cohort A1: Non-metastatic/ Resectable (with planned or you are undergoing therapy)- your cancer has not spread, may be able to remove it with operation
  Interventions: Other: Non-Metastatic and Resectable
- Metastatic and Un-resectable: Cohort A2: Metastatic/ Unresectable (with planned or you are undergoing therapy)- your cancer has spread, not able to operate at this time to take out all the cancer
  Interventions: Other: Metastatic and Un-resectable
- No evidence of disease, under surveillance: Cohort B: No evidence of disease/ surveillance (you have completed initial therapy)- currently there is no evidence of your cancer/disease and you are under surveillance, meaning your physician is checking your medical situation at intervals or occasionally for any sign of changes
  Interventions: Other: No evidence of disease, under surveillance
- ALT or WDLS: Cohort C: You have been diagnosed with ALT (atypical lipoma) or WDLS (well-differentiated liposarcoma)
  Interventions: Other: ALT or WDLS

INTERVENTIONS:
Other: Non-Metastatic and Resectable — Blood Draw Timepoints:
  * Before any treatment begins
  * After Neo-adjuvant therapy (only if you receive this type of therapy)
  * After local surgery
  * After Adjuvant therapy (only if you receive this type of therapy)
  * Follow up after adjuvant therapy: at Months 3, 6, 9, 12, 15, 18, and 24
  * After evidence of recurrence or worsening of disease, and then collected at standard of care disease evaluation visits up until 24 months from the last treatment for the initial diagnosis
  Groups: Non-Metastatic and Resectable
Other: Metastatic and Un-resectable — Blood Draw Timepoints:
  * Before any treatment begins
  * During standard of care disease evaluation visits for up to 24 months
  Groups: Metastatic and Un-resectable
Other: No evidence of disease, under surveillance — Blood Draw Timepoints:
  * From completion of treatment- at Months 3, 6, 9, 12, 15, 18, and 24; depending on when you enroll into the study you will start at the next timepoint in this schedule
  * After evidence of recurrence or worsening of disease, and then collected at standard of care disease evaluation visits up until 24 months from the last treatment for the initial diagnosis
  Groups: No evidence of disease, under surveillance
Other: ALT or WDLS — Blood Draw Timepoints:
  • Collect once after surgery (up to six weeks after surgery)
  Groups: ALT or WDLS

SUMMARY:
The purpose of this research study is to see how well Low Pass Whole Genome Sequencing (LP-WGS) can detect circulating tumor deoxyribonucleic acid (ctDNA) in the blood of participants who have bone or soft tissue sarcoma (type of cancer).

DETAILED DESCRIPTION:
In this ever-expanding age of precision oncology, the stagnant treatment algorithms and subsequent oncologic outcomes for sarcoma patients highlight the need for novel technologies to help clinicians treat these patients. While countless prognostic and therapeutic molecular biomarkers have been identified for many other cancers, sarcoma practitioners have strikingly few tumor markers to guide treatment. The development of a sarcoma-specific liquid biopsy could greatly help clinicians with diagnosis, prognostication, treatment response, minimal recurrent disease, and recurrence. The purpose of this study is to clinically evaluate ctDNA liquid biopsy approaches in adult and pediatric patients with bone and soft tissue sarcomas.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent or assent when applicable from the participant, LAR, parent or legal guardian and HIPAA authorization for release of personal health information.
2. All ages allowed
3. Suspected or confirmed disease (must meet one of the criteria below):

   1. Suspected bone or soft tissue tumor concerning for sarcoma (pending confirmation of sarcoma diagnosis)

      OR
   2. Suspected lipomatous mass concerning for ALT or WDLS with planned surgery

      OR
   3. Confirmed bone or soft tissue sarcoma meeting one of the criteria below:

      * Non-metastatic/Resectable sarcoma with either planned or currently receiving therapy
      * Metastatic or unresectable sarcoma, with planned or currently receiving therapy
      * Non-metastatic sarcoma under surveillance with no more than 1 year from completion of therapy

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages with concern for or diagnosed with bone or soft tissue sarcoma or lipomatous mass will be identified by treatment investigators in oncology clinics treatment patients with sarcoma
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with ctDNA detected | Approximately 24 months
  A binary variable indicating whether or not ctDNA was detected by low pass whole genome sequencing (LP-WGS) in the sample.

SECONDARY OUTCOMES:
Quantity of ctDNA detected | Approximately 24 months
  A longitudinal continuous variable indicating the quantitative levels of ctDNA in the sample as measured by LP-WGS. Timepoints include pre-treatment, at disease evaluations during treatment, post-treatment, at remission/complete response (if applicable), during surveillance (if applicable), and at recurrence/progression (if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Johann Hsu, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina